CLINICAL TRIAL: NCT04849858
Title: Pilot Study of Liposomal Bupivacaine Redosing in Patients Undergoing Major Gynecologic Procedures: A Quality Improvement Project in Post-operative Pain
Brief Title: Pilot Study of Liposomal Bupivacaine Redosing in Patients Undergoing Major Gynecologic Procedures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jill Tseng, Assistant Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20194981; UCI 19-16 (Other: UCI CFCCC)
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Fibroids; Uterine Cancer
Keywords: ovarian cancer; fibroids; uterine cancer; Transverse abdominis plane block; TAP block
MeSH Terms: conditions — Ovarian Neoplasms; Leiomyoma; Uterine Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study with retrospective data analysis. Patients will be assigned to treatment groups on a consecutive basis. We will be recruiting 45 eligible patients from our University of California Irvine (UCI) gynecologic oncology clinic. Each clinic patient who is scheduled for surgery will be screened for eligibility. The first 15 patients enrolled will receive perioperative plain bupivacaine transversus abdominis plane (TAP) blocks. The next 15 patients enrolled will receive perioperative single-dose Liposomal Bupivacaine (LB) TAP blocks. The final 15 patients enrolled will receive perioperative LB TAP blocks followed by redosing of the TAP blocks in 48-60 hours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bupivacaine TAP Block (Active Comparator): The first 15 patients enrolled will receive perioperative plain bupivacaine TAP blocks.
  Interventions: Drug: Bupivacaine
- Liposomal Bupivacaine TAP Block (Active Comparator): After enrolling all 15 participants in the first arm, the next 15 patients enrolled will receive perioperative single-dose Liposomal Bupivacaine TAP blocks.
  Interventions: Drug: Liposomal bupivacaine
- Liposomal Bupivacaine TAP Block with Re-dosing (Active Comparator): After enrolling all 30 patients in the first two arms, the final 15 patients enrolled will receive perioperative Liposomal Bupivacaine TAP blocks followed by redosing of the TAP blocks in 48-60 hours.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Participants in this group will receive a TAP block using the drug Bupivacaine.
  Arms: Bupivacaine TAP Block
Drug: Liposomal bupivacaine — Participants in this group will receive a TAP block using the drug Liposomal Bupivacaine.
  Arms: Liposomal Bupivacaine TAP Block
Drug: Liposomal bupivacaine — Participants in this group will receive a TAP block using the drug Liposomal Bupivacaine followed by a re-dosing during their hospitalization
  Other Names: With Re-dosing
  Arms: Liposomal Bupivacaine TAP Block with Re-dosing

SUMMARY:
The purpose of this research study is to find out which type of transversus abdomens plane (TAP) and block (bupivacaine, liposomal bupivacaine or liposomal bupivacaine with re-dosing at 48-60 hours) improves your pain control and lowers your risk of post-operative common side effects of surgery and narcotic pain medications.

DETAILED DESCRIPTION:
The purpose of this research study is to find out which type of TAP block (bupivacaine, liposomal bupivacaine or liposomal bupivacaine with re-dosing at 48-60 hours) improves your pain control and lowers your risk of post-operative common side effects of surgery and narcotic pain medications.

An anesthesiologist participating on this study will describe the TAP block to you during your preoperative interview and will obtain your consent for the block procedure with your anesthesia consent prior to the procedure. TAP blocks are one of the various methods of controlling your pain after surgery. They are typically placed with an anesthetic agent, such as bupivacaine. The U.S. Food and Drug Administration (FDA) has recently approved a longer-acting form of the anesthetic used in this study, liposomal bupivacaine. Although both medications, bupivacaine and liposomal bupivacaine are approved by the FDA, there are only a few trials such as this one, in the United States, comparing the various types of TAP blocks. No studies exist comparing the re-dosing of a TAP block, as we will be doing in this study.

Currently, the standard of care after a gynecologic procedure may or may not include receiving a TAP block. This was a decision typically made, with your consent, at the discretion of an anesthesiologist and your surgeon. As per the standard of care, after surgery, you would be given oral pain medications to control your pain and intravenous pain medications for severe breakthrough pain. Our study will not change your post-operative pain medication schedule or timing. It will only study the effectiveness of the TAP block you get in controlling your pain.

Even though the medicines (bupivacaine or liposomal bupivacaine) used in this study are FDA-approved, the use of these drugs in this study is investigational.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years old
* Must be undergoing an open gynecologic procedure through a midline vertical incision with a gynecologic oncologist

Exclusion Criteria

* History of chronic pain
* History of opioid dependence
* Suspected or confirmed history of endometriosis
* History of fibromyalgia
* Suspected or confirmed interstitial cystitis or painful bladder syndrome
* History of or current opioid use prior to surgery
* Hypersensitivity to bupivacaine
* Severe hepatic or renal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study applies to patients receiving care with a gynecologic oncologist
Enrollment: 13 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid consumption | Post-operative day 0 to day 8
  Morphine equivalents (milligrams)

SECONDARY OUTCOMES:
Pain at rest and during activity | Post-operative day 0 to day 8
  Measured pain on a Visual Analog Scale (VAS), Scale 0 (no pain) - 10 (high pain)
Nausea/Vomiting | Post-operative day 0 to day 8
  Presence or Absence of nausea or vomiting
Ileus | Post-operative day 0 to day 8
  Presence or Absence of Ileus
Bowel Function | Post-operative day 0 to day 8
  Time to return of bowel function (days)
Ambulation | Post-operative day 0 to day 8
  Time to first ambulation (days)
Hospital stay | Post-operative day 0 to day 8
  Length of hospital stay (days)
Surgical Adverse Events | Post-operative day 0 to day 8
  Presence or Absence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jill H Tseng, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No